CLINICAL TRIAL: NCT07119775
Title: Tideglusib: Expanded Access Use in Congenital Myotonic Dystrophy
Status: Available | Type: Expanded Access
Sponsor: AMO Pharma Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: AMO-02 Expanded Access
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Congenital Myotonic Dystrophy
Keywords: Tideglusib; Congenital Myotonic Dystrophy; Myotonic Dystrophy; Dystrophia Myotonica; Myotonia Atrophica; Myotonia Dystrophica; Myotonic Dystrophy, Congenital Steinert Disease; Steinert Myotonic Dystrophy; Steinert's Disease
MeSH Terms: conditions — Myotonic Dystrophy | interventions — tideglusib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tideglusib

SUMMARY:
This treatment plan is limited to a single patient with Congenital Myotonic Dystrophy, who is ineligible or otherwise unable to participate in ongoing clinical trials.

Age Groups: Child, Adult, Older Adult